CLINICAL TRIAL: NCT04864899
Title: Clinical Significance of Subclinical Myocardial Involvement in Recovered COVID-19 Patients Using Cardiovascular Magnetic Resonance (R-COVID-CMR)
Acronym: R-COVID-CMR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Ng Ming-Yen, Clinical Assistant Professor, The University of Hong Kong
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: UW21-005
Record Dates: First submitted 2021-03-19; First posted 2021-04-29 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2025-05

CONDITIONS: Covid19; Viral Respiratory Infection
MeSH Terms: conditions — COVID-19 | interventions — Hematologic Tests; Walk Test

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Recovered COVID-19 patients (Experimental)
  Interventions: Diagnostic Test: Cardiac Magnetic Resonance Imaging (CMR); Diagnostic Test: Blood test; Diagnostic Test: 6-minute walk test
- Recovered non-COVID-19 viral respiratory infections patients (Experimental)
  Interventions: Diagnostic Test: Cardiac Magnetic Resonance Imaging (CMR); Diagnostic Test: Blood test; Diagnostic Test: 6-minute walk test
- Age and gender matched controls (Experimental)
  Interventions: Diagnostic Test: Cardiac Magnetic Resonance Imaging (CMR); Diagnostic Test: Blood test; Diagnostic Test: 6-minute walk test

INTERVENTIONS:
Diagnostic Test: Cardiac Magnetic Resonance Imaging (CMR) — Imaging
Diagnostic Test: Blood test — Blood investigation
Diagnostic Test: 6-minute walk test — Correlating the cardiac MRI parameters with functional capacity

SUMMARY:
This is a prospective cohort study that aims to clinical significance of subclinical myocardial involvement in recovered COVID-19 patients using cardiovascular magnetic resonance.

DETAILED DESCRIPTION:
This study aims to:

1. Determine the extent of myocardial involvement of COVID-19, as assessed by Cardiovascular Magnetic Resonance (CMR), 2 weeks after patient recovery, at 3-month post discharge and at 1-year post discharge.
2. Correlate these myocardial characteristics to biventricular structure, function, blood biomarkers of inflammation, clinical symptoms, and functional capacity at all time points.
3. Follow up recovered COVID-19 patients beyond the end of this study to assess for hard outcomes such as death, heart failure hospitalization, cardiac arrest and ventricular tachycardia/ fibrillation.

Recovered COVID-19 patients and age and gender matched controls subjects will be recruited.

ELIGIBILITY:
Inclusion Criteria:

• Recovered COVID-19 patients

Definition of recovered COVID-19 patient:

* COVID-19 diagnosis = established by a positive reverse transcription polymerase chain reaction (RT-PCR) for severe acute respiratory syndrome coronavirus-2 [SARS-CoV2] and recovered from COVID-19.
* Recovery = based on two criteria: (1) two negative nasopharyngeal swab RT-PCR results >24 hours apart and (2) absence of fever and improvement in respiratory symptoms.

  * Recovered non-COVID-19 patients with viral respiratory infections confirmed with viral polymerase chain reaction testing AND with a confirmed negative COVID-19 RT-PCR test.
  * Age and gender matched controls with no cardiac risk factors, not on cardiac medications, no history of myocardial infarction, heart failure or myocarditis, negative COVID-19 RT-PCR test and negative COVID-19 antibodies test.

Exclusion Criteria:

* Previous myocardial infarction or myocarditis unrelated to COVID-19 infection
* History of heart failure unrelated to COVID-19 infection
* Presence of pacemakers or implantable cardiac defibrillators
* Any contraindication for CMR testing
* Renal impairment with eGFR <45ml/min/1.73m2
* Limited life expectancy <1 year, for example due to pulmonary disease, cancer or significant hepatic failure
* Refusal or inability to sign an informed consent.
* Potential for non-compliance towards the requirements in the trial protocol (especially the medical treatment) or follow-up visits

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2024-08-06 (Actual); Study Completion 2024-08-06 (Actual)

PRIMARY OUTCOMES:
The extent of myocardial involvement, as assessed by CMR tissue characterisation (T1/ T2/ ECV/ LGE), change from 2 weeks after patient recovery, at 3-months post discharge and at 1-year post discharge. | 2 years
The correlation of these myocardial characteristics to biventricular structure at all time-points. | 2 years
The correlation of these myocardial characteristics to biventricular function (CMR cine/strain) at all time-points. | 2 years
The correlation of these myocardial characteristics to blood biomarkers of inflammation at all time-points. | 2 years
The correlation of these myocardial characteristics to clinical symptoms at all time-points. | 2 years
The correlation of these myocardial characteristics to functional capacity (6 minute walk test) at all time-points. | 2 years

SECONDARY OUTCOMES:
Follow-up patients beyond the end of this study to assess for hard outcomes such as death. | 2 years
Follow-up patients beyond the end of this study to assess for hard outcomes such as heart failure hospitalisation. | 2 years
Follow-up patients beyond the end of this study to assess for hard outcomes such as cardiac arrest. | 2 years
Follow-up patients beyond the end of this study to assess for hard outcomes such as ventricular tachycardia/ fibrillation. | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- The University of Hong Kong, Hong Kong, Hong Kong